CLINICAL TRIAL: NCT01527032
Title: Risk-adapted Therapy for AL Amyloidosis
Brief Title: Risk-adapted Therapy for Primary Systemic (AL) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2174
Record Dates: First submitted 2011-07-28; First posted 2012-02-06 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-07

CONDITIONS: Amyloidosis
Keywords: amyloidosis; stem cell transplant
MeSH Terms: conditions — Amyloidosis | interventions — Melphalan; Thalidomide; Dexamethasone

INTERVENTIONS:
Drug: melphalan, thalidomide and dexamethasone

SUMMARY:
High-dose melphalan (MEL) with autologous stem cell transplant (SCT) is an effective therapy for systemic AL amyloidosis (AL), but treatment-related mortality (TRM) has historically been high. The investigators performed a phase II trial of risk-adapted SCT followed by adjuvant dexamethasone (dex) and thalidomide (thal) in an attempt to reduce TRM and improve response rates. Patients with newly diagnosed AL involving £2 organ systems were assigned to MEL 100, 140, or 200 mg/m2 with SCT, based on age, renal function and cardiac involvement. Patients with persistent clonal plasma cell disease 3 months post-SCT received 9 months of adjuvant thal/dex (or dex if there was a history of deep vein thrombosis or neuropathy). TRM was 4.4%. Thirty-one patients began adjuvant therapy, with 16 (52%) completing 9 months of treatment and 13 (42%) achieving an improvement in hematological response. By intention-to-treat, overall hematological response rate was 71% (36% complete response) with 44% having organ responses. With a median follow-up of 31 months, 2-year survival was 84% (95% confidence interval: 73%, 94%). Risk-adapted SCT with adjuvant thal/ dex is feasible and results in low TRM and high hematological and organ response rates in AL patients.

DETAILED DESCRIPTION:
High-dose melphalan (MEL) with autologous stem cell transplant (SCT) is an effective therapy for systemic AL amyloidosis (AL), but treatment-related mortality (TRM) has historically been high. The investigators performed a phase II trial of risk-adapted SCT followed by adjuvant dexamethasone (dex) and thalidomide (thal) in an attempt to reduce TRM and improve response rates. Patients (n=45) with newly diagnosed AL involving £2 organ systems were assigned to MEL 100, 140, or 200 mg/m2 with SCT, based on age, renal function and cardiac involvement. Patients with persistent clonal plasma cell disease 3 months post-SCT received 9 months of adjuvant thal/dex (or dex if there was a history of deep vein thrombosis or neuropathy). Organ involvement was kidney (67%), heart (24%), liver/GI (22%) and peripheral nervous system (18%), with 31% having two organs involved. TRM was 4.4%. Thirty-one patients began adjuvant therapy, with 16 (52%) completing 9 months of treatment and 13 (42%) achieving an improvement in hematological response. By intention-to-treat, overall hematological response rate was 71% (36% complete response) with 44% having organ responses. With a median follow-up of 31 months, 2-year survival was 84% (95% confidence interval: 73%, 94%). Risk-adapted SCT with adjuvant thal/ dex is feasible and results in low TRM and high hematological and organ response rates in AL patients.(British Journal of Haematology 2007;139:224-33)

Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Study Completion 2005-09 (Actual)